CLINICAL TRIAL: NCT00513617
Title: Arginine Supplementation in Sickle Cell Anemia: Physiological and Prophylactic Effects
Brief Title: Effectiveness of Arginine as a Treatment for Sickle Cell Anemia
Acronym: Arginine
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UCSF Benioff Children's Hospital Oakland (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Lori Styles/Principal Investigator, Childrens Hospital of Oakland and Research Institute
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 485; U54HL070587-04 (NIH)
Record Dates: First submitted 2007-08-06; First posted 2007-08-08 (Estimated); Results first posted 2009-08-04 (Estimated); Last update posted 2017-03-29 (Actual); Status verified 2009-06

CONDITIONS: Anemia, Sickle Cell
Keywords: Sickle Cell Disease; Anemia; Nitric Oxide; Vaso Occlusive Events; Arginine Supplementation
MeSH Terms: conditions — Anemia, Sickle Cell; Anemia; Vaso-Occlusive Crises | interventions — Arginine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Low Dose (Active Comparator): 0.05 g/kg/day Arginine
  Interventions: Drug: Arginine
- High Dose (Active Comparator): 0.10 g/kg/day Arginine
  Interventions: Drug: Arginine
- Placebo (Placebo Comparator): No Arginine
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Arginine — Depending on the weight of the child or adult, the patients took any where between 4-10 capsules 2 times a day. Patients weighing less than 45 kilograms were on the low dose active (or placebo) so the capsules were smaller. Patients greater than or equal to 45 kgs were on the high dose active or placebo, so these capsules were larger.
  Arms: High Dose; Low Dose
Drug: Placebo — Depending on the weight of the child or adult, the patients took any where between 4-10 capsules 2 times a day. Patients weighing less than 45 kilograms were on the low dose active (or placebo) so the capsules were smaller. Patients greater than or equal to 45 kgs were on the high dose active or placebo, so these capsules were larger.
  Arms: Placebo

SUMMARY:
Sickle cell disease (SCD), also known as sickle cell anemia, is an inherited genetic disease that can cause intense pain episodes. This study will evaluate the effectiveness of the nutritional supplement arginine at improving blood cell function and disease symptoms in people with SCD.

DETAILED DESCRIPTION:
SCD is an inherited blood disorder. Symptoms include anemia, infections, organ damage, and intense episodes of pain that are called "sickle cell crises." SCD is caused by an abnormal type of hemoglobin, which is a protein inside red blood cells that carries oxygen. In people with SCD, the abnormal hemoglobin distorts the shape of the red blood cells. This causes the red blood cells to clump together, decreasing blood flow and oxygen delivery to the body's tissues. The reduced levels of oxygen can lead to sickle cell crises and tissue damage. Hemolysis, the destruction of red blood cells, is also a hallmark of SCD. During hemolysis, hemoglobin is released into the bloodstream, where it removes nitric oxide (NO), a natural chemical in the body that expands blood vessels. Arginase, another protein released during hemolysis, removes arginine from the bloodstream, which can also lead to decreased NO levels. The lack of NO constricts blood vessels, further contributing to painful sickle cell crises. Arginine supplementation may increase healthy hemoglobin and NO production and, in turn, prevent or reduce sickle cell crises. The purpose of this study is to evaluate the effectiveness of arginine at increasing NO levels, improving red blood cell function, and reducing hospitalizations and pain medication use in people with SCD.

This study will enroll children and adults with SCD. Participants will be randomly assigned to receive twice daily doses of either a low dose of arginine, a high dose of arginine, or placebo for 12 weeks. Study visits will occur at baseline, three times during Month 1, and Weeks 8, 12, 14, and 16. Each study visit will include an echocardiogram to measure heart activity, blood collection, and a medical history review to identify adverse events, pain medication usage, headaches, emergency department visits, and hospitalizations.

ELIGIBILITY:
Inclusion Criteria:

* Established diagnosis of H SS or S-beta thalassemia
* History of at least one vaso-occlusive pain event in the 12 months prior to study entry
* Regular compliance with comprehensive medical care
* In a steady disease state and not in the midst of any acute complication due to SCD at study entry

Exclusion Criteria:

* Inability to take or tolerate oral medications
* Liver dysfunction (i.e., SGPT level greater than or equal to two times the normal limit and albumin level less than or equal to 3.2 g/dL)
* Kidney dysfunction ( i.e., creatinine level greater than or equal to 1.2 mg/dL for children and greater than or equal to 1.4 mg/dL for adults)
* Allergy to arginine
* Pregnant
* Received a blood transfusion within the 90 days prior to study entry
* More than 10 hospital admissions for pain in the 12 months prior to study entry
* Daily use of opioids and experiencing unstable pain that interferes with work or daily routine
* Required more than 3 hospital admissions and more than 10 emergency department/day hospital visits in the 12 months prior to study entry
* Received treatment with hydroxyurea within the 90 days prior to study entry
* Received treatment with any investigational drug in the 90 days prior to study entry

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2004-06; Primary Completion 2007-09 (Actual); Study Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lillian McMahon, MD, Principal Investigator — Boston Medical Center; Rathi Iyer, MD, Principal Investigator — University of Mississippi Medical Center (Pediatric); Carolyn Bigelow, MD, Principal Investigator — University of Mississippi Medical Center (Adult); Lennette Benjamin, MD, Principal Investigator — Montefiore Medical Center; Mary Fabry, MD, Principal Investigator — Albert Einstein College of Medicine; Thomas Moulton, MD, Principal Investigator — Children's Hospital of Montefiore; Kim Smith-Whitley, MD, Principal Investigator — Children's Hospital of Philadelphia; Laura DeCastro, MD, Principal Investigator — Duke University; Kenneth Ataga, MD, Principal Investigator — University of North Carolina, Chapel Hill; Samir K. Ballas, MD, Principal Investigator — Thomas Jefferson University; Sal Bertalone, MD, Principal Investigator — Kosair Children's Hospital; Carlton Dampier, MD, Principal Investigator — St. Christopher's Childrens Hospital; William Mentzer, MD, Principal Investigator — University of California, San Francisco; Winfred Wang, MD, Principal Investigator — St. Jude's Childrens Research Hospital; Ulrike Reiss, MD, Principal Investigator — St. Jude Children's Research Hospital; Cynthia Rutherford, MD, Principal Investigator — Children's Medical Center Dallas; Kathryn Hassell, MD, Principal Investigator — University of Colorado, Denver; Joan Parkhurst Cain, MD, Principal Investigator — Children's Hospital of Oklahoma
Locations (17):
- United States (17):
  - Children's Hospital of Oakland and Research Institute, Oakland, California
  - University of California - San Francisco, San Francisco, California
  - University of Colorado at Denver and Health Sciences Center--Sickle Cell Treatment and Research Center, Denver, Colorado
  - Kosair Children's Hospital, Louisville, Kentucky
  - Boston Medical Center, Boston, Massachusetts
  - University of Mississippi Medical Center (Adult), Jackson, Mississippi
  - University of Mississippi Medical Center (Pediatric), Jackson, Mississippi
  - Montefiore Medical Center, The Bronx, New York
  - Children's Hospital of Montefiore, The Bronx, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Children's Hospital of Oklahoma, Oklahoma City, Oklahoma
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - St. Christopher's Children's Research Hospital, Philadelphia, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - Children's Medical Center of Dallas, Dallas, Texas

REFERENCES:
- [Derived] Bolarinwa AB, Oduwole O, Okebe J, Ogbenna AA, Otokiti OE, Olatinwo AT. Antioxidant supplementation for sickle cell disease. Cochrane Database Syst Rev. 2024 May 22;5(5):CD013590. doi: 10.1002/14651858.CD013590.pub2. PMID 38775255

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrolled subjects at participating sites from May 2004 through July 2007. Sites consisted of sickle cell treatment centers from across the United States.
Pre-assignment Details: All subjects were to be without hydroxyurea, transfusion, and arginine for 90 days prior to enrollment. Prior to randomization, blood was drawn for baseline efficacy and safety measurements.
Groups:
- Low Dose: 0.05 g/kg/day of Arginine in capsule form
- High Dose: 0.10 g/kg/day of Arginine in capsule form
Period: Overall Study
Arm/Group | Low Dose | High Dose | Placebo
Started | 36 | 35 | 38
Completed | 25 | 25 | 30
Not Completed | 11 | 10 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Low Dose | High Dose | Placebo | Total
Number analyzed (Participants) | 36 | 35 | 38 | 109
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 14 | 18 | 18 | 50
  Between 18 and 65 years | 22 | 17 | 20 | 59
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 24.5 (12.85) | 20.0 (10.01) | 21.0 (11.49) | 23.2 (11.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 19 | 20 | 60
  Male | 15 | 16 | 18 | 49
Region of Enrollment [Number; unit: participants]
  United States | 36 | 35 | 38 | 109.0
Genotype of SCD [Number; unit: participants]
  Sickle cell S-Beta Thalassemia (SB0) | 2 | 3 | 2 | 7.0
  Sickle cell Anemia (SS) | 34 | 32 | 36 | 102.0

OUTCOME MEASURES:

1. Primary Outcome: Gardos Channel Activity
Description: Gardos channel activity: a calcium (Ca2+)-activated K+ channel
Time Frame: 12 weeks after randomization
Population: All subjects that were randomized and dosed - Intent to Treat (ITT) No imputation used.
Measure: Mean (Standard Deviation); unit: mmol/10^13 cells x min
Arm/Group | Low Dose | High Dose | Placebo
Number analyzed (Participants) | 12 | 11 | 14
mmol/10^13 cells x min | -0.0342 (0.2341) | 0.0043 (0.3028) | 0.1076 (0.2822)
Statistical Analysis 1: Comparison: Low Dose vs Placebo; Null hypothesis is no difference between high vs. placebo and low vs. placebo in change from baseline at Week 12 post-randomization. Separate models were fit for pediatric and adult populations, however the combined population is entered here; Test type: Superiority or Other; p = 0.080, Mixed Models Analysis — Alpha was set at 0.05; Null is tested using the F-test from a random effects longitudinal mixed model, with treatment and baseline measurement as fixed effects; Mean Difference (Final Values) = -0.1254, Standard Error of Mean 0.0705 — Placebo was subtracted from the Low dose
Statistical Analysis 2: Comparison: High Dose vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.133, Mixed Models Analysis — Alpha was set at 0.05; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.0980, Standard Error of Mean 0.0713 — Placebo was subtracted from High dose

2. Secondary Outcome: Soluble Vascular Cell Adhesion Molecule
Description: Soluble vascular cell adhesion molecule (sVCAM) a vascular adhesion molecule
Time Frame: 12 weeks after randomization
Reporting Status: Not Posted

3. Primary Outcome: Nitric Oxide
Description: Nitric oxide from plasma amino acids
Time Frame: 12 weeks after randomization
Population: All subjects that were randomized and dosed - ITT No imputation used.
Measure: Mean (Standard Deviation); unit: uM
Arm/Group | Low Dose | High Dose | Placebo
Number analyzed (Participants) | 12 | 11 | 14
uM | -3.8697 (15.7574) | 2.9250 (11.1646) | -3.0265 (18.6887)
Statistical Analysis 1: Comparison: Low Dose vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.915, Mixed Models Analysis — Alpha was set at 0.5; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.1826, Standard Error of Mean 0.0713 — Placebo subtracted from Low dose
Statistical Analysis 2: Comparison: High Dose vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.918, Mixed Models Analysis — Alpha was set at 0.05; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 2.3582, Standard Error of Mean 4.1047 — Placebo subtracted from High dose

4. Primary Outcome: Mean Corpuscular Hemoglobin Concentration
Description: Mean corpuscular hemoglobin concentration as measured by an Advia machine
Time Frame: 12 weeks after randomization
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Low Dose | High Dose | Placebo
Number analyzed (Participants) | 12 | 11 | 14
g/dL | -1.8485 (6.3092) | 0.7692 (2.2165) | -0.0705 (1.4422)
Statistical Analysis 1: Comparison: Low Dose vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.015, Mixed Models Analysis — Alpha was set at 0.05; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -1.7867, Standard Error of Mean 1.1101 — Placebo subtracted from Low dose
Statistical Analysis 2: Comparison: High Dose vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.557, Mixed Models Analysis — Alpha was set at 0.05; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.5213, Standard Error of Mean 1.1553 — Placebo subtracted from High dose

5. Secondary Outcome: 8-iso-PGF2a
Description: 8-iso-PGF2a is a measure of lipid peroxidation and oxidative damage in vivo measured by enzyme immunoassay kit from Cayman chemical
Time Frame: 12 weeks after randomization
Reporting Status: Not Posted

6. Secondary Outcome: Endothelin-1
Description: Endothelin-1 is a potent vasoconstrictor and pro-inflammatory agent which is elevated in SCD patients
Time Frame: 12 weeks after randomization
Reporting Status: Not Posted

7. Secondary Outcome: Fetal Hemoglobin
Description: Fetal hemoglobin (HbF) as measured by the Advia machine
Time Frame: 12 weeks after randomization
Reporting Status: Not Posted

LIMITATIONS AND CAVEATS:
Adult enrollment was slower than expected. Adult subjects were more likely than peds to drop-out due to SCD pain crisis. Higher doses of arginine (such as used in animal studies) were limited by number of daily pills required.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No